CLINICAL TRIAL: NCT01176812
Title: Dermal Filling Agents: Patient Satisfaction
Brief Title: Dermal Fillers Patient Satisfaction
Status: Withdrawn | Type: Observational
Why Stopped: Difficult to recruit subjects in the area.
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: 9251
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2011-02

CONDITIONS: Loss of Facial Fat
Keywords: Facialwasting; Juvederm; Restylane

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dermal Fillers: Facial Wasting

SUMMARY:
The face is arguably the most critical aesthetic unit of the body. As humans begin to age, numerous changes occur to the face. Changes include the formation of wrinkles, soft-tissue atrophy, gravitational descent resulting in sagging skin, loss of skin and muscle tone, and changes in bony architecture. These changes are potentiated in our population secondary to sun exposure and smoking. To combat the effects of aging on the face, a multitude of products and procedures exist to attempt to reverse the effects of sun damage and aging to achieve a youthful and rejuvenated appearance. There has been a shift from invasive procedures such as a facelift to noninvasive means using filling agents to restore lost contour deformities.

The investigators hypothesis is that the use of dermal filling agents effectively delays the need for invasive procedures such as facelifts, and that patient satisfaction has increased with the evolution of recent dermal filling agents.

DETAILED DESCRIPTION:
The first part of this study will involve a retrospective review of patients who have had a dermal filler injection between 01/01/1998 through 12/31/2008 and then following up with one (1) patient satisfaction survey. The first part of the study, which is retrospective, may involve approximately 500 subjects. The data collected from the retrospective review will be the subject's name, medical record number, and address for contact information. Any other data collected will come from the answers on the questionnaire.

The second part of this study will be a prospective study involving 100 subjects who are scheduled to have a dermal filler injection. These subjects will be asked to complete one (1) patient satisfaction survey two weeks after injection. Facial photos will be taken before the injection and then two weeks after injection at the follow up visit. This will complete the subject's participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from 21 - 80 years of age who are scheduled to have a dermal filler injection.

Exclusion Criteria:

* Subjects under 21 years of age or older than 80 years of age will be excluded from this study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have an interest in combating the effects of facial aging with injectible dermal fillers.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Satisfaction with results of dermal filler | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R David, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States